CLINICAL TRIAL: NCT02182427
Title: Malnutrition Clinical Characteristics Validation Study
Acronym: MCC
Status: Completed | Type: Observational
Sponsor: Academy of Nutrition and Dietetics (Other)
Collaborators: American Society for Parenteral and Enteral Nutrition (Other)
Responsible Party: Principal Investigator, Alison Steiber, Chief Science Officer, Academy of Nutrition and Dietetics
Other Study IDs: 2014-Pilot
Record Dates: First submitted 2014-07-01; First posted 2014-07-08 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No

SUMMARY:
Malnutrition (under-nutrition) occurs in approximately 30% of hospitalized adults worldwide and results in poor outcomes. However there is no universal method for diagnosing malnutrition. A group of experts created a set of 6 characteristics to identify malnutrition. The goal of this project is to determine whether these characteristics are the best indicators to identify malnutrition or if there are other factors that may better identify malnutrition. Because there is no gold standard definition for malnutrition, the investigators will compare the characteristics against outcomes such as length of stay, hospital readmission and death. Outcomes are also influenced by disease state, therefore, information on what brought the patient to the hospital and what happened to them in the hospital will be collected that allows the investigators to separate the effect of malnutrition from disease. The hypothesis for this study is that the malnutrition clinical characteristics and diagnosis criteria, as presented by the experts, are valid and reliable principles for the diagnosis of adult under-nutrition.

ELIGIBILITY:
Inclusion Criteria:

* Patient on inpatient dietitian consult list
* Able to speak English to answer questions
* Ability to provide informed consent (or provided by family member)
* Expected remaining admission time > 24 hours (determined by no mention of pending discharge in physicians notes)
* Age ≥ 18 years

Exclusion Criteria:

* Seen previously by Registered Dietitian during current admission
* Patient on hospice or palliative care, in a psychiatric, maternity, pediatric or day surgery area, or in dedicated trauma or burn unit.
* Life expectancy <7 days per physician note or Registered Dietitian (RD) judgment
* Participated in the study during a previous admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All eligible patients (according to the inclusion and exclusion criteria seen below) who are admitted to one of the following acute care facilities: University Hospitals Case Medical Center, Cleveland Clinic, and St. John's Westshore in Cleveland, Ohio, United States, and Princess Alexandra Hospital in Brisbane, Queensland, Australia.
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2014-04; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Number of participants diagnosed with and without malnutrition using the MCC. | 30-days post-discharge

SECONDARY OUTCOMES:
30-day readmission rate among study participants | Within 90 days after data collection is complete

CONTACTS AND LOCATIONS:
Overall Officials: Alison Steiber, Principal Investigator — Academy of Nutrition and Dietetics; Maree Ferguson, Study Chair — Princess Alexandra Hospital
Locations (4):
- United States (3):
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - St. John's West Shore Hospital, Westlake, Ohio
- Princess Alexandra Hospital, Brisbane, Queensland, Australia

REFERENCES:
- [Background] White JV, Guenter P, Jensen G, Malone A, Schofield M; Academy of Nutrition and Dietetics Malnutrition Work Group; A.S.P.E.N. Malnutrition Task Force; A.S.P.E.N. Board of Directors. Consensus statement of the Academy of Nutrition and Dietetics/American Society for Parenteral and Enteral Nutrition: characteristics recommended for the identification and documentation of adult malnutrition (undernutrition). J Acad Nutr Diet. 2012 May;112(5):730-8. doi: 10.1016/j.jand.2012.03.012. Epub 2012 Apr 25. PMID 22709779